CLINICAL TRIAL: NCT01652417
Title: Randomized, Multicentric Study Evaluating the Efficacy and the Safety of Methylprednisolone Bolus in the Treatment of Renal Sarcoidosis
Brief Title: Treatment of Renal Sarcoidosis by Methylprednisolone Bolus
Acronym: CORTICOIDOSE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient recruitment
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P 110118; AOM 11003 (Other: Assistance Publique)
Record Dates: First submitted 2012-05-16; First posted 2012-07-30 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2015-10

CONDITIONS: Renal Sarcoidosis
Keywords: Methylprednisolone; prednisone; renal sarcoidosis treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- oral prednisone (No Intervention): Oral prednisone 1 mg/kg/d for 30 days and progressive tapering of steroids, to get 0,5 mg/kg/d at M3 and 0,25 mg/kg/d at M6 and 5-10 mg at M12.
- methylprednisolone bolus (Experimental): methylprednisolone bolus 15 mg/kg/d for 3 days before oral prednisone 1 mg/kg/d for 30 days and progressive tapering of steroids, to get 0,5 mg/kg/d at M3 and 0,25 mg/kg/d at M6 and 5-10 mg at M12.
  Interventions: Drug: methylprednisolone bolus IV 15 mg/kg/d for 3 days.

INTERVENTIONS:
Drug: methylprednisolone bolus IV 15 mg/kg/d for 3 days. — methylprednisolone bolus IV 15 mg/kg/d for 3 days.
  Other Names: Methylprenisolone Mylan
  Arms: methylprednisolone bolus

SUMMARY:
Renal sarcoidosis treatment is based on steroids, but the dose and duration are unknown. Despite this treatment, most patients will have chronic kidney disease. From our previous studies, the investigators believe that high dose steroids by methylprednisolone bolus will improve patient outcome and renal function.

DETAILED DESCRIPTION:
In a multicentric, randomized, open trial, the investigators will assess the efficacy of methylprednisolone bolus at 15mg/kg/d for 3 days before oral steroids on renal function improvement in renal sarcoidosis patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Acute kidney injury with estimated glomerular filtration rate (eGFR) < 60 mL/min/1,73 m2, defined by an increase of initial value > 25% or an increase of > 30 µmol/l, since at least 3 months.
* Sarcoidosis diagnostic criteria according to ATS/ERS/WASOG (Am J Respir Crit Care Med 1999)
* Renal biopsy compatible with renal sarcoidosis :
* Granulomatosis tubulo-interstitial nephropathy and extra-renal damage of histologically proved or suggestive sarcoidosis Or
* Tubulo-interstitial nephropathy without granuloma and extra-renal damage of histologically proved sarcoidosis
* Informed consent
* Patients with social security

Exclusion Criteria:

* Corticosteroids greater than 0,25 mg/kg/j prednisone equivalent
* Introduction of an immunosuppressant in the month before inclusion
* Another cause of renal granulomatosis or tubulo-interstitial nephropathy
* Isolated renal damage without extra-renal past or present damage for a sarcoidosis
* Chronic renal failure, prior sarcoidosis with eGFR < 30 mL/min/1,73 m2
* Acute renal failure from other causes. If hypercalcaemia is greater than 3 mmol/L, the correction of any dehydration will systematically salt intake, followed of renal function control before inclusion.
* Pregnancy, nursing
* Tuberculosis
* Uncontrolled sepsis
* Uncontrolled psychotic state
* Hypersensibility to methylprednisolone hemisuccinate
* Drugs prescription causing wave burst arrhythmia and/or long QT on ECG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-10; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with a positive response defined by eGRF better than 100% compared to eGRF prior treatment or a normalization of renal function. | 3 months after the beginning of the treatment

SECONDARY OUTCOMES:
Efficacy (eGFR, percentage of patients with a eGRF < 60 ml/min/1.73m²) | 1, 3, 6 and 12 months after the beginning of the treatment
Extra-renal manifestations | 1, 3, 6 and 12 months after the beginning of the treatment
incidence of arrhythmias and cardiac conduction disease | 1, 3, 6 and 12 months after the beginning of the treatment
fragility fracture | 1, 3, 6 and 12 months after the beginning of the treatment
neuro-psychiatric troubles and infections | 1, 3, 6 and 12 months after the beginning of the treatment
number of renal and extra-renal relapses. | 1, 3, 6 and 12 months after the beginning of the treatment
Characterization of vitamin and calcium deficiencies by blood and urinary dosages | 1, 3, 6 and 12 months after the beginning of the treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Néphrologie et Dialyses, Hôpital Tenon, Paris, France

REFERENCES:
- [Derived] Mahevas M, Audard V, Rousseau A, Cez A, Guerrot D, Verhelst D, Delahousse M, Hanrotel C, Pillebout E, Daugas E, Krastinova E, Valeyre D, Boffa JJ; GSF French Sarcoidosis Group. Efficacy and safety of methylprednisolone pulse followed by oral prednisone vs. oral prednisone alone in sarcoidosis tubulointerstitial nephritis: a randomized, open-label, controlled clinical trial. Nephrol Dial Transplant. 2023 Mar 31;38(4):961-968. doi: 10.1093/ndt/gfac227. PMID 36066903